CLINICAL TRIAL: NCT03058419
Title: An Open-label Drug Interaction Study in Healthy Subjects to Evaluate the Effect of Oral Doses of JNJ-54175446 on the Inhibition of Cytochrome P450 CYP3A4, CYP2C9, CYP1A2 and CYP2D6 Activity and the Induction of CYP2B6 and CYP2C19 Activity Using a Multiple Probe Substrate Cocktail
Brief Title: A Study to Evaluate the Effect of Oral Doses of JNJ-54175446 on the Inhibition of Cytochrome P450 CYP3A4, CYP2C9, CYP1A2 and CYP2D6 Activity and the Induction of CYP2B6 and CYP2C19 Activity Using a Multiple Probe Substrate Cocktail in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108283; 2016-004167-39 (EudraCT Number); 54175446EDI1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-02-16; First posted 2017-02-20 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-54175446; Midazolam; Warfarin; Caffeine; Dextromethorphan; Bupropion; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug Cocktail + JNJ-54175446 (Experimental): All subjects will receive a single dose of drug cocktail (consisting of midazolam [2 milligram (mg)], warfarin [10 mg], caffeine [50 mg], dextromethorphan [30 mg], bupropion [150 mg] and omeprazole [20 mg]) on Day 1, 7 and 11; JNJ-54175446 150 mg on Day 7, 9, 10 and 11 and JNJ-54175446 600 mg on Day 8.
  Interventions: Drug: JNJ-54175446 150 mg; Drug: JNJ-54175446 600 mg; Drug: Midazolam 2 mg; Drug: Warfarin 10 mg; Drug: Caffeine 50 mg; Drug: Dextromethorphan 30 mg; Drug: Bupropion 150 mg; Drug: Omeprazole 20 mg

INTERVENTIONS:
Drug: JNJ-54175446 150 mg — Subjects will receive JNJ-54175446 150 mg capsules orally (1*100 mg + 1*50 mg) under fasted conditions on Day 7, 9, 10 and 11.
Drug: JNJ-54175446 600 mg — Subjects will receive JNJ-54175446 600 mg (6*100 mg capsules) orally on Day 8.
Drug: Midazolam 2 mg — Subjects will receive midazolam 2 mg oral emulsion [2 (milligram per milliliter (mg/mL)] as a drug cocktail on Day 1, 7 and 11.
Drug: Warfarin 10 mg — Subjects will receive warfarin 10 mg tablets (2*5 mg) orally as a drug cocktail on Day 1, 7 and 11.
Drug: Caffeine 50 mg — Subjects will receive caffeine 50 mg tablet (1*50 mg) orally as a drug cocktail on Day 1, 7 and 11.
Drug: Dextromethorphan 30 mg — Subjects will receive dextromethorphan 30 mg capsule (1*30 mg) orally as a drug cocktail on Day 1, 7 and 11.
Drug: Bupropion 150 mg — Subjects will receive Bupropion 150 mg tablet (1*150 mg) orally as a drug cocktail on Day 1, 7 and 11.
Drug: Omeprazole 20 mg — Subjects will receive omeprazole 20 mg capsule (1*20 mg) orally as a drug cocktail on Day 1, 7 and 11.

SUMMARY:
The main purpose of this study is to determine the potential inhibitory/inducing effects of JNJ-54175446 after single and repeated dosing on the single-dose pharmacokinetics (PK) of a cocktail, containing selective probes of cytochrome P450 (CYP) enzymes (CYP3A4/A5, CYP2C9, CYP1A2, CYP2D6, CYP2B6, and CYP2C19) in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2), inclusive (BMI = weight/height^2)
* Subject must be healthy on the basis of physical examination, medical history, vital signs, and triplicate 12-lead electrocardiograms (ECGs), including QTc according to Fridericia's formula (QTcF) less than or equal to (</=) 450 milliseconds (ms) for males and </= 470 ms for females, performed at screening and first admission to the study site
* Subject must be healthy on the basis of clinical laboratory tests performed at screening and Day -1. If the results of the hematology, serology, serum chemistry (excluding liver function tests, which must be in normal range of 1.25 * upper limit of normal laboratory range), and coagulation panel, or urinalysis are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities to be not clinically significant
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, a male subject: Who is sexually active with a woman of childbearing potential and has not had vasectomy must agree to use a barrier method of contraception (eg, condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository). In addition, their female partner should also use a highly effective method of birth control (example, hormonal contraception) for at least the same duration. Who is sexually active with a woman who is pregnant must use a condom and Must agree not to donate sperm
* A female subject must be of non-childbearing potential at screening

Exclusion Criteria:

* Subject has a history of or current liver or renal insufficiency (estimated creatinine clearance below 60 milliliter per minute (mL/min), significant skin disease such as, but not limited to, dermatitis, eczema, Stevens-Johnson Syndrome, drug rash, psoriasis or urticaria, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic (including coagulation disorders), rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness that the investigator considers should exclude the subject
* Subject has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening
* Subject has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening
* Subject has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that, in the opinion of the investigator, with written concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)
* Subject has a history of drug or alcohol use disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria within 6 months before screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 17
  The Cmax is the maximum observed plasma concentration.
Plasma Trough Concentration (Ctrough) | Up to Day 17
  Ctrough is defined as observed plasma concentration of drug just prior to the beginning or at the end of a dosing interval.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Day 17
  The Tmax is defined as actual sampling time to reach maximum observed concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC [0-Last]) | Up to Day 17
  The AUClast is the area under the plasma concentration-time curve from time zero to the time of the last measurable (non-below quantification limit) concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Up to Day 17
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda [z]) | Up to Day 17
  Lambda (z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) | Up to Day 17
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Apparent Total Clearance (CL/F) | Up to Day 17
  Apparent total clearance is calculated as dose/AUC(0-infinity).
Apparent Volume of Distribution (Vd/F) | Up to Day 17
  Apparent volume of distribution, calculated as dose/(lambda[z]*AUC[0-infinity]).
Parent to Metabolite Ratio (Cmax) | Up to Day 17
  Parent to metabolite ratio Cmax is defined as the ratio of individual Cmax values between parent and metabolite.
Parent to Metabolite Ratio (AUC [Last]) | Up to Day 17
  Parent to metabolite ratio (AUC [Last]) is defined as ratio of individual (AUC [Last]) values between parent and metabolite.
Parent to Metabolite Ratio (AUC [infinity]) | Up to Day 17
  Parent to Metabolite Ratio (AUC [infinity]) is defined as the ratio of individual (AUC [infinity]) values between parent and metabolite.

SECONDARY OUTCOMES:
Number of Subjects With Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to follow up (14 to 21 days after last dose)
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium